CLINICAL TRIAL: NCT07059663
Title: Synergic Effects of Schroth Method With and Without Core Stabilization Exercises in Idiopathic Scoliosis Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Lahore (Other)
Responsible Party: Principal Investigator, Faiza Sarwar, Physical Therapist, University of Lahore
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Faiza.sarwar
Record Dates: First submitted 2025-07-01; First posted 2025-07-11 (Actual); Last update posted 2025-07-15 (Actual); Status verified 2025-07

CONDITIONS: Scoliosis; Scoliosis Idiopathic
Keywords: Schroth Method; Idiopathic Scoliois; Core Stabilization Exercises; Cobb Angle; Lumbar Extensor Endurance; Chest mobility; SRS-22 questionnaire; Postural correction; Spinal deformity; Physiotherapy
MeSH Terms: conditions — Scoliosis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Schroth method with Core Stabilization Exercises (Experimental): The Schroth method and core stabilization exercises will be performed three times a week for 10 weeks, with each session lasting 60 minutes
  Interventions: Other: Schroth Method with Core Stabilization Exercises
- Schroth Method (Active Comparator): this group will receive the core stabilization exercises alone
  Interventions: Other: Schroth Method

INTERVENTIONS:
Other: Schroth Method with Core Stabilization Exercises — The Schroth method will focus on postural correction techniques aimed at improving spinal alignment, reducing the curvature of the spine, and enhancing trunk control. Key exercises will include spinal elongation, de-rotation, and specific breathing techniques to help reduce the scoliotic curve. Core stabilization exercises will target the deep trunk muscles, such as the transversus abdominis and multifidus, to improve spinal stability. These exercises will involve bodyweight exercises, resistance bands, and stability balls, aimed at increasing muscle endurance and promoting better posture. The interventions will be performed three times a week for 10 weeks, with each session lasting 60 minutes
  Arms: Schroth method with Core Stabilization Exercises
Other: Schroth Method — The control group will receive the Schroth method alone, focusing solely on postural correction exercises. These exercises will aim to improve spinal alignment, reduce curvature, and enhance postural control through spinal elongation, de-rotation, and specific breathing techniques designed to address the scoliosis. The control group will not receive any core stabilization exercises in addition to the Schroth method. This intervention will also be performed three times a week for 10 weeks, with each session lasting 60 minutes
  Arms: Schroth Method

SUMMARY:
A randomized controlled trial was conducted on 72 patients diagnosed with idiopathic scoliosis at the University of Lahore Teaching Hospital. The study aimed to explore the synergistic effects of the Schroth method with and without core stabilization exercises. Participants were randomly allocated into two groups: Group A, which received both the Schroth method and core stabilization exercises, and Group B, which received only the Schroth method. The intervention lasted for 10 weeks, with assessments conducted at baseline, the 5th week, and the 10th week. Outcome measures included Cobb angle (spinal curvature), lumbar extensor endurance (Sorensen test), chest mobility, and quality of life (SRS-22 questionnaire). The study found significant improvements in all outcome measures for both groups, with Group A showing superior results. The addition of core stabilization exercises to the Schroth method resulted in better reductions in Cobb angle, enhanced lumbar extensor endurance, and improved chest mobility and quality of life, indicating a synergistic effect of the combined approach. The findings suggest that incorporating core stabilization exercises into scoliosis treatment protocols can lead to superior clinical outcomes.

DETAILED DESCRIPTION:
A randomized controlled trial will be conducted at the University of Lahore Teaching Hospital. Thirty patients diagnosed with idiopathic scoliosis, aged 10 to 18 years, will be randomly divided into two groups: Group A will receive the Schroth method in combination with core stabilization exercises, while Group B will receive only the Schroth method. Both interventions will be delivered three times weekly for ten weeks. Outcome measures, including Cobb angle (curve magnitude), lumbar extensor endurance (Sorensen test), chest mobility, and quality of life (SRS-22), will be assessed at baseline, week 5, and week 10.

ELIGIBILITY:
Inclusion Criteria:

* • Age 10 to 18

  * X-ray diagnosed of idiopathic scoliosis with Cobb Angle 10˚- 30˚
  * Participants with Idiopathic Scoliosis
  * Both genders will be included
  * Scoliosis with Down syndrome.

Exclusion Criteria:

* Any neurological condition such as cerebral palsy or epilepsy.
* Any other orthopedic condition such as hip dysplasia, osteogenesis imperfecta, or leg length discrepancy.
* Surgical history of the spine, such as spinal fusion and decompression surgery.
* Severe systemic disorders such as autoimmune disorders, severe cardiovascular conditions
* Non-Idiopathic Scoliosis

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 72 (Estimated)
Dates: Start 2025-07-30 (Estimated); Primary Completion 2025-09-10 (Estimated); Study Completion 2026-01-30 (Estimated)

PRIMARY OUTCOMES:
Change in Cobb Angle(Curve Magnitude) | Change from Pre-Intervention to the 10th week
  The Cobb angle will be used to measure the reduction in spinal curvature. The Cobb angle is the standard method for assessing the severity of scoliosis. A decrease in the Cobb angle indicates improvement in spinal alignment
Change in Lumbar Extensor Endurance (Sorensen Test) | Change from pre-intervention to 10th week
  The Sorensen test will assess lumbar extensor muscle endurance, measuring the ability to hold an isometric contraction for as long as possible. Improvements in endurance indicate better trunk stability
Change in Chest Mobility (measured by chest expansion) | Change from pre-intervention to 10th week
  Chest mobility will be measured using a non-stretch measuring tape at the xiphoid level, both at rest and during maximal inhalation and exhalation. An increase in chest mobility is an indicator of improved thoracic flexibility and lung function.
Change in Quality of Life (SRS-22 Questionnaire) | Change from pre-intervention to 10th week
  The Scoliosis Research Society (SRS-22) questionnaire will be used to assess the quality of life, including function, pain, mental health, self-image, and satisfaction with treatment. Improvements in scores reflect enhanced functional outcomes and psychosocial well-being. Each item is rated on a 5-point Likert scale (1 = worst, 5 = best).
  Total score ranges from 22 to 110. Higher scores indicate better quality of life and treatment satisfaction.

CONTACTS AND LOCATIONS:
Locations (1):
- UOL Teaching Hospital, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: Undecided
Can only be requested from principal investigator

REFERENCES:
- [Background] Kocaman H, Bek N, Kaya MH, Buyukturan B, Yetis M, Buyukturan O. The effectiveness of two different exercise approaches in adolescent idiopathic scoliosis: A single-blind, randomized-controlled trial. PLoS One. 2021 Apr 15;16(4):e0249492. doi: 10.1371/journal.pone.0249492. eCollection 2021. PMID 33857180
- [Background] Egea-Gamez RM, Galan-Olleros M, Martinez-Caballero I, Ramirez-Barragan A, Serrano JI, Palazon-Quevedo A, Gonzalez-Diaz R. Scoliosis in Adolescent Patients With Down Syndrome: Correlation Between Curve Magnitude and Functional Level. Clin Spine Surg. 2023 Dec 1;36(10):E471-E477. doi: 10.1097/BSD.0000000000001495. Epub 2023 Jul 14. PMID 37448188
- [Background] Day JM, Fletcher J, Coghlan M, Ravine T. Review of scoliosis-specific exercise methods used to correct adolescent idiopathic scoliosis. Arch Physiother. 2019 Aug 23;9:8. doi: 10.1186/s40945-019-0060-9. eCollection 2019. PMID 31463082
- [Background] Ceballos-Laita L, Carrasco-Uribarren A, Cabanillas-Barea S, Perez-Guillen S, Pardos-Aguilella P, Jimenez Del Barrio S. The effectiveness of Schroth method in Cobb angle, quality of life and trunk rotation angle in adolescent idiopathic scoliosis: a systematic review and meta-analysis. Eur J Phys Rehabil Med. 2023 Apr;59(2):228-236. doi: 10.23736/S1973-9087.23.07654-2. Epub 2023 Jan 24. PMID 36692412